## The Effects of Motor Imagery Training and Physical Practice on Upper Extremity Motor Function in Patients with Stroke

NCT05526612 09/02/2022

## **Statistical Analysis**

The conformity of the variables to the normal distribution in each group will be analyzed with the Shapiro-Wilk test. Descriptive statistics for the variables conforming to the normal distribution will be given as mean±standard deviation (minimum-maximum). For discrete and non-normal distribution variables, descriptive statistics will be given as median (1st quartile-3 quartile).

Intra-group variation will be analyzed with Paired Samples t-test for continuous variables, and Wilcoxon Signed Rank test for discrete and non-normally distributed variables. In the comparison between groups, change values will be calculated as "percentage change [(after treatment-before treatment)/before treatment x 100]" for all variables.

Comparison of the groups will be made with Independent Samples t-test for variables conforming to normal distribution, Mann Whitney-U test for discrete and non-normally distributed variables, and Chi-square test for categorical variables. In analyzes based on SPSS, p<0.05 will be considered statistically significant.

G\*Power Ver.3.0.10 program was used to calculate the sample size in the study. In order for the study to have a power of 85% with a margin of error of 0.05, a total of 32 individuals, 16 individuals in both groups, will be included in the study.

In the study, 32 stroke patients will be divided into 2 separate groups, in which physical practice of motor imagery to be done with Bobath Therapeutic Approach (BTA+MI) and physical practice of imagery activities to be done with Bobath Therapeutic Approach after motor imagery (BTA+MI+PP) will be performed using a computer-based program before evaluation, via www.randomizer.org site.

## **Informed Consent Form**

## Dear volunteer,

Before deciding whether or not to participate in this research, you need to know why and how the research will be conducted. Therefore, it is very important to read and understand this form. Take the time to carefully read the information below. If you wish, discuss this information with your family and/or relatives. If there is something that you do not understand and is not clear to you, or if you want more information, ask the researcher.

We invite you to a research titled "The Effects of Motor Imagery Training and Physical Practice on Upper Extremity Motor Function in Stroke Patients". The aim of this study, led by Prof.Dr. Arzu Razak ÖZDİNÇLER and co-researcher Nisa Nur SOYSAL, is to examine the effects of specific functional task-oriented motor imagery training combined with the Bobath Therapeutic Approach and post-imagery physical practice on eating activity and upper extremity motor function in stroke patients.

You are invited to this study because you have a diagnosis of stroke. You are requested to participate in our study for an average of 50 minutes, 2 days a week, for a total of 8 weeks. In our study, 32 participants will be randomly divided into 2 groups with you. The first group in the treatment program; Motor imagery (BTA+MI) to be done with the Bobath Therapeutic Approach and physical practice of the imagery activities (BTA+MI+PP) after the motor imagery to be done with the second group Bobath Therapeutic Approach will be done. Motor imagery activity was determined as 'eating activity'. Before and after the treatment, we need to fill out some evaluation forms and videotape you.

The treatment program to be applied in this study will not harm you. You should know that we will be careful not to share your information and video recording with a third party who is not involved in the study. At the same time, your information will never be shared with third parties unless you agree. Your medical and identity information will be kept confidential and your identity information will not be disclosed even if the research is published. You should know that you will not make any payment or receive any payment for participating in this study. At the same time, no fee will be charged from you or the social security institution you are affiliated with for the evaluations provided to you within the study.

Participation in this study is completely voluntary. You have the right not to participate in the study or to leave at any stage. In order to reach the right conclusion in the study, you are expected to give the most appropriate answers while answering the questions in the evaluation forms, without being under pressure or indoctrination from anyone. The information obtained from these forms will be used for research purposes only.

| Under these conditions, I agree to participate in the research in question voluntarily, without any pressure or suggestion. |
|---|
| Name and Surname of the Participant/Guardian/Guardian: |
| Signature/Date: |
| Name and Surname of Person Witnessing Consent: |
| Signature/Date: |
| Principal Investigator Name and Surname: |
| Signature: |